CLINICAL TRIAL: NCT00925652
Title: ABCDE: A Phase II Randomized Study of Adjuvant Bevacizumab, Metronomic Chemotherapy (CM), Diet and Exercise After Preoperative Chemotherapy for Breast Cancer
Brief Title: Bevacizumab, Metronomic Chemotherapy (CM), Diet and Exercise After Preoperative Chemotherapy for Breast Cancer
Acronym: ABCDE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated early due to slow accrual.
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Beth Israel Deaconess Medical Center (Other); Translational Breast Cancer Research Consortium (Other); Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Erica Mayer, MD, MPH, Erica Mayer, M.D., Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-134; AVF 4571s; TBCRC 012
Record Dates: First submitted 2009-06-19; First posted 2009-06-22 (Estimated); Results first posted 2022-01-19 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2021-12

CONDITIONS: Breast Cancer
Keywords: CM; bevacizumab; cyclophosphamide; methotrexate; exercise intervention; diet intervention
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; Cyclophosphamide; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Lifestyle: Diet (Experimental): The dietary intervention focuses on the Food Pyramid, emphasizing diet that is low in fat and high in fruits, vegetables and fiber. Patients receive a series of 13 telephone calls over the course of one-year with a dedicated and trained counselor.
  Interventions: Behavioral: Lifestyle: Diet
- Lifestyle: Diet+Exericise (Experimental): The dietary intervention focuses on the Food Pyramid, emphasizing diet that is low in fat and high in fruits, vegetables and fiber. The exercise intervention is comprised of a target physical activity goal of 180 minutes of moderate-intensity activity each week. Patients receive a series of 13 telephone calls over the course of one-year with a dedicated and trained counselor.
  Interventions: Behavioral: Lifestyle: Diet; Behavioral: Lifestyle: Diet+Exercise
- Lifestyle: Diet and Bevicizumab+CM (Experimental): The dietary intervention focuses on the Food Pyramid, emphasizing diet that is low in fat and high in fruits, vegetables and fiber. Patients receive a series of 13 telephone calls over the course of one-year with a dedicated and trained counselor.
  Bevicizumab: 15 mg/kg administered intravenously day 1 of a 3-week cycle for 6 months and day 1 of a 6 week cycle up to 2 years Cyclophosphamide: 50 mg orally each day of a 3-week cycle for 6 months Methotrexate: 2.5 mg orally twice daily of a 3-week cycle for 6 months
  Interventions: Drug: Bevacizumab; Drug: Cyclophosphamide; Drug: Methotrexate; Behavioral: Lifestyle: Diet
- Lifestyle: Diet+Exericise and Bevicizumab+CM (Experimental): The dietary intervention focuses on the Food Pyramid, emphasizing diet that is low in fat and high in fruits, vegetables and fiber. The exercise intervention is comprised of a target physical activity goal of 180 minutes of moderate-intensity activity each week. Patients receive a series of 13 telephone calls over the course of one-year with a dedicated and trained counselor.
  Bevicizumab: 15 mg/kg administered intravenously day 1 of a 3-week cycle for 6 months and day 1 of a 6 week cycle up to 2 years Cyclophosphamide: 50 mg orally each day of a 3-week cycle for 6 months Methotrexate: 2.5 mg orally twice daily of a 3-week cycle for 6 months
  Interventions: Drug: Bevacizumab; Drug: Cyclophosphamide; Drug: Methotrexate; Behavioral: Lifestyle: Diet; Behavioral: Lifestyle: Diet+Exercise

INTERVENTIONS:
Drug: Bevacizumab
  Other Names: Avastin
  Arms: Lifestyle: Diet and Bevicizumab+CM; Lifestyle: Diet+Exericise and Bevicizumab+CM
Drug: Cyclophosphamide
  Other Names: Cytoxan
  Arms: Lifestyle: Diet and Bevicizumab+CM; Lifestyle: Diet+Exericise and Bevicizumab+CM
Drug: Methotrexate
  Other Names: MTX
  Arms: Lifestyle: Diet and Bevicizumab+CM; Lifestyle: Diet+Exericise and Bevicizumab+CM
Behavioral: Lifestyle: Diet
Behavioral: Lifestyle: Diet+Exercise
  Arms: Lifestyle: Diet+Exericise; Lifestyle: Diet+Exericise and Bevicizumab+CM

SUMMARY:
If residual breast cancer is found in the breast or lymph node tissue removed after preoperative chemotherapy, one may be at increased risk of breast cancer recurrence in the future. The purpose of this research study is to determine if having additional treatment after preoperative chemotherapy and surgery with bevacizumab and metronomic chemotherapy would make a difference in reducing the participants chance of breast cancer recurrence compared to the standard of care, which is observation alone. This study will also evaluate the potential additional benefits from participating in an exercise and dietary intervention compared to the dietary intervention alone. Because no one knows which which post-neoadjuvant strategy is best, participants will be "randomized" to one of the study groups: 1. Diet Intervention arm, 2. Diet and Exercise Intervention Arm, 3. Bevacizumab, cyclophosphamide, methotrexate and diet intervention, 4. Bevacizumab, cyclophosphamide, methotrexate, diet and exercise intervention arm.

DETAILED DESCRIPTION:
Bevacizumab is an antibody that is made in the laboratory. Bevacizumab works differently from the way chemotherapy drugs work. Bevacizumab works to slow or stop the growth of cells in cancer tumors by decreasing the blood supply to tumors. Bevacizumab has been approved by the U.S Food and Drug Administration to treat advanced colorectal, lung and kidney cancers. Metronomic chemotherapy also attacks tumor blood supply. Standard chemotherapy drugs are used, cyclophosphamide and methotrexate (CM), but in very small daily doses by mouth, well below the threshold where they can cause people to feel sick. Previous research studies have shown that women with breast cancer who take metronomic CM and bevacizumab feel very well, and the combination therapy is active in reducing their cancer. Participants in this study will also be provided with diet or diet and exercise counseling over the telephone. Studies have shown that many women who are treated for breast cancer will gain weight during and after their treatment, and may also experience fatigue and weakness. Many studies have shown that making changes in diet and increasing exercise can help prevent weight gain and also may increase energy and decrease other side effects of chemotherapy and other breast cancer treatments.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed invasive breast cancer. HER2 positive disease is not allowed. Metastatic breast cancer (Stage IV) is not allowed.
* For patients entering the trial after neoadjuvant chemotherapy, there must be the presence of residual invasive disease on pathologic review following neoadjuvant chemotherapy. Residual disease is defined as a Miller-Payne response in the breast of 0-4 and/or residual carcinoma in one or more regional lymph nodes that would meet AJCC 7th edition criteria for N1 - N3 disease. The presence of DCIS without invasion does not qualify as residual disease. Alternatively, if Miller-Payne grading is not available, the patient will be eligible if the pathology report indicates any residual invasive carcinoma following neoadjuvant therapy.
* If tumor is triple negative (ER-/PR-/HER2-) and the patient received neoadjuvant chemotherapy, disease may be clinical stage I-III pre-operatively, per AJCC 7th edition, based on baseline evaluation by clinical examination and/or breast imaging. Patients must have the presence of residual invasive disease on pathologic review following their neoadjuvant chemotherapy.
* If tumor is triple negative and the patient did not receive neoadjuvant chemotherapy, there must be pathologic lymph node positivity and Stage IIB or greater disease after surgery. For the purposes of eligibility, lymph node positivity can refer to either axillary or intramammary lymph nodes.
* If tumor is hormone receptor positive, disease must be clinical Stage III neoadjuvantly, per AJCC 7th edition, based on baseline evaluation by clinical examination and/or breast imaging, or pathologic Stage IIB or greater at time of definitive surgery. Patients with hormone receptor positive breast cancer who do not receive neoadjuvant chemotherapy are not eligible for this protocol.
* For patients who completed neoadjuvant chemotherapy, the regimen must contain an anthracycline, a taxane, or both. Patients who have received neoadjuvant therapy as part of a clinical trial are acceptable. Protocol therapy must be initiated < 180 days after last surgery for breast cancer. For triple negative patients who receive adjuvant chemotherapy only, the regimen must contain both an anthracycline and a taxane. For these patients, protocol therapy must be initiated < 28 weeks after initiation of adjuvant chemotherapy.
* Patients with ER+ and/or PR+ breast cancer should receive adjuvant hormonal therapy
* No prior exposure to bevacizumab or other inhibitors of angiogenesis is allowed.
* Patients must have completed definitive resection of primary tumor. Negative margins for both invasive and ductal carcinoma in situ (DCIS) are desirable, however positive margins are acceptable if the treatment team believes no further surgery is possible and patient has received radiotherapy. Patients with margins positive for lobular carcinoma in situ are eligible.
* Post-mastectomy radiotherapy is suggested for all patients with a primary tumor 5cm or greater or involvement of 4 or more lymph nodes. Whole breast radiotherapy is required for patients who underwent breast conserving therapy, including lumpectomy, partial mastectomy, and excisional biopsy.
* Patients must have the presence of residual invasive disease on pathologic review following their preoperative chemotherapy. The presence of DCIS without invasion does not qualify as residual disease. Alternatively, if Miller-Payne grading is not available, the patient will be eligible if the pathology report indicates any residual invasive carcinoma following preoperative therapy.
* LVEF equal to or greater than institutional limits of normal after preoperative chemotherapy, as assessed by echocardiogram, within 30 days prior to registration
* ECOG Performance Status 0-1 within 2 weeks of registration
* 18 years of age or greater

Exclusion Criteria:

* Laboratory assessments as outlined in the protocol
* Stage IV breast cancer. Patients with metastatic disease are ineligible. However, specific staging studies are not required in the absence of symptoms
* Prior history of hypertensive crisis or hypertensive encephalopathy
* History if myocardial infarction or unstable angina within 12 months prior to registration
* History of stroke or transient ischemic attack at any time
* Significant vascular disease within 6 months prior to registration
* History of hemoptysis within 1 month prior to registration
* Ongoing or active infection
* NYHA Grade II or greater congestive heart failure
* Unstable angina pectoralis
* Psychiatric illness/social situations that would limit compliance with study requirements
* Evidence of bleeding diathesis or significant coagulopathy
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to registration or anticipation of need for major surgical procedure during the course of the study
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to registration
* History of abdominal fistula or gastrointestinal perforation within 6 months prior to registration
* Serious, non-healing wound, active ulcer, or unhealed bone fracture
* Known hypersensitivity to any component of bevacizumab or compounds of similar chemical or biologic composition to cyclophosphamide or methotrexate
* Known HIV infection, as immunosuppression could be worsened by use of cyclophosphamide and methotrexate, and the impact of chemotherapy and/or bevacizumab therapy on the pharmacology of standard anti-HIV therapy is not known
* Patient may not be pregnant, expect to become pregnant, plan to conceive a child while on study or breastfeeding.
* Prior history of any malignancy treated without curative intent, or treated with curative intent within the past 5 years. Prior history of DCIS > 5 years before current breast cancer diagnosis is acceptable if ipsilateral (and no radiotherapy given) or contralateral (with or without radiotherapy) or contralateral (with or without radiotherapy). Prior history of contralateral stage 1 breast cancer > 5 years prior to the current breast cancer diagnosis is acceptable, however prior ER/PR+ breast cancer > stage 1 at any time is not allowed.
* Patients with a pleural effusion or abdominal ascites are excluded because of the theoretical risk for methotrexate accumulation and related toxicity
* Current use of anticoagulants is allowed as long as patients have been on a stable dose for more than two weeks with stable INR
* Chronic therapy with full dose aspirin or standard non-steroidal anti-inflammatory agents is allowed
* While on study, patients may not receive other investigational agents as part of other clinical trials
* Adjuvant bisphosphonate use, on or off of clinical trial, is allowed. Patients may be started on adjuvant bisphosphonate therapy either before or after ABCDE trial enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2015-01-30 (Actual); Study Completion 2019-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erica Mayer, MD, Study Chair — Dana-Farber Cancer Institute
Locations (9):
- United States (9):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Indiana Unversity Simon Cancer Center, Indianapolis, Indiana
  - Faulkner Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at Milford Regional Medical Center, Milford, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of North Carolina Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Trapani D, Jin Q, Miller KD, Rugo HS, Reeder-Hayes KE, Traina T, Abdou Y, Falkson C, Abramson V, Ligibel J, Chen W, Come S, Nohria A, Ryabin N, Tayob N, Tolaney SM, Burstein HJ, Mayer EL. Optimizing Postneoadjuvant Treatment of Residual Breast Cancer With Adjuvant Bevacizumab Alone, With Metronomic or Standard-Dose Chemotherapy: A Combined Analysis of DFCI 05-055 and DFCI 09-134/TBCRC 012/ABCDE Clinical Trials. Clin Breast Cancer. 2025 Jun;25(4):e419-e430.e5. doi: 10.1016/j.clbc.2024.12.018. Epub 2024 Dec 31. PMID 39890560

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lifestyle: Diet | Lifestyle: Diet+Exericise | Lifestyle: Diet and Bevicizumab+CM | Lifestyle: Diet+Exericise and Bevicizumab+CM
Started | 13 | 13 | 11 | 13
Withdraw | 6 | 5 | 3 | 1
Off Treatment Because of Other Complicating Disease | 0 | 0 | 2 | 3
Off Treatment Because of Disease Recurrence | 1 | 3 | 0 | 0
Lost of Follow-up | 0 | 1 | 0 | 0
Death | 0 | 0 | 0 | 3
Completed | 6 | 4 | 6 | 6
Not Completed | 7 | 9 | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lifestyle: Diet | Lifestyle: Diet+Exericise | Lifestyle: Diet and Bevicizumab+CM | Lifestyle: Diet+Exericise and Bevicizumab+CM | Total
Number analyzed (Participants) | 13 | 13 | 11 | 13 | 50
Age, Continuous [Median (Full Range); unit: years] | 48 [36 to 64] | 43 [34 to 56] | 57 [25 to 63] | 48 [31 to 63] | 47.5 [25 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 11 | 13 | 49
  Male | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 11 | 13 | 50

OUTCOME MEASURES:

1. Primary Outcome: Median 3-year Recurrence-free Survival (RFS)
Description: RFS events is defined as the duration of time from randomization to time of an RFS event, marked as positive if any of listed event shows: local failure (invasive), regional failure, distant failure, contralateral breast cancer (invasive), any other second cancer (excluding non-melanomatous skin cancer or cervical cancer in situ), or death from any cause. The diagnosis of local or distant recurrence should be pathologically confirmed however if biopsy if not possible, radiology confirmation acceptable.
Time Frame: Disease assessments occurred every 12 weeks on treatment and every 6 months in long-term follow-up up to 7.5 years.
Measure: Median (95% Confidence Interval); unit: years
Groups:
- Lifestyle: Diet: The dietary intervention focuses on the Food Pyramid, emphasizing diet that is low in fat and high in fruits, vegetables and fiber. Patients receive a series of 13 telephone calls over the course of one-year with a dedicated and trained counselor.
  Lifestyle: Diet
- Lifestyle: Diet+Exericise: The dietary intervention focuses on the Food Pyramid, emphasizing diet that is low in fat and high in fruits, vegetables and fiber. The exercise intervention is comprised of a target physical activity goal of 180 minutes of moderate-intensity activity each week. Patients receive a series of 13 telephone calls over the course of one-year with a dedicated and trained counselor.
  Lifestyle: Diet
  Lifestyle: Diet+Exercise
- Lifestyle: Diet and Bevicizumab+CM: The dietary intervention focuses on the Food Pyramid, emphasizing diet that is low in fat and high in fruits, vegetables and fiber. Patients receive a series of 13 telephone calls over the course of one-year with a dedicated and trained counselor.
  Bevicizumab: 15 mg/kg administered intravenously day 1 of a 3-week cycle for 6 months and day 1 of a 6 week cycle up to 2 years Cyclophosphamide: 50 mg orally each day of a 3-week cycle for 6 months Methotrexate: 2.5 mg orally twice daily of a 3-week cycle for 6 months
  Bevacizumab
  Cyclophosphamide
  Methotrexate
  Lifestyle: Diet
- Lifestyle: Diet+Exericise and Bevicizumab+CM: The dietary intervention focuses on the Food Pyramid, emphasizing diet that is low in fat and high in fruits, vegetables and fiber. The exercise intervention is comprised of a target physical activity goal of 180 minutes of moderate-intensity activity each week. Patients receive a series of 13 telephone calls over the course of one-year with a dedicated and trained counselor.
  Bevicizumab: 15 mg/kg administered intravenously day 1 of a 3-week cycle for 6 months and day 1 of a 6 week cycle up to 2 years Cyclophosphamide: 50 mg orally each day of a 3-week cycle for 6 months Methotrexate: 2.5 mg orally twice daily of a 3-week cycle for 6 months
  Bevacizumab
  Cyclophosphamide
  Methotrexate
  Lifestyle: Diet
  Lifestyle: Diet+Exercise
Arm/Group | Lifestyle: Diet | Lifestyle: Diet+Exericise | Lifestyle: Diet and Bevicizumab+CM | Lifestyle: Diet+Exericise and Bevicizumab+CM
Number analyzed (Participants) | 13 | 13 | 11 | 13
years | 0.68 [0.44 to 1] | 0.5 [0.24 to 1] | 0.86 [0.63 to 1] | 0.2 [0.04 to 1]

2. Secondary Outcome: Feasibility Rate
Description: The feasibility of post-adjuvant maintenance metronomic chemotherapy is open to women with hormone receptor negative tumors and either node negative or node positive disease.
Time Frame: 2 years
Population: data not collected
Arm/Group | Lifestyle: Diet | Lifestyle: Diet+Exericise | Lifestyle: Diet and Bevicizumab+CM | Lifestyle: Diet+Exericise and Bevicizumab+CM
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Number of Serious Adverse Event of Bevacizumab
Description: Adverse event evaluations will occur at each study visit throughout the treatment period of 2 years and will continue every 6 months during the follow-up period. Only Grade 3/4 AE (CTCAE v4) was reported.
Time Frame: Followed every 6 months for 7.5 years after study entry, or completion of final analysis, whichever comes first.
Measure: Number; unit: cases
Arm/Group | Lifestyle: Diet and Bevicizumab+CM | Lifestyle: Diet+Exericise and Bevicizumab+CM
Number analyzed (Participants) | 11 | 13
cases | 12 | 8

4. Secondary Outcome: Number of Serious Adverse Event of Metronomic Chemotherapy
Description: as for outcome 3
Time Frame: Followed every 6 months for 7.5 years after study entry, or completion of final analysis, whichever comes first.
Measure: Number; unit: cases
Arm/Group | Lifestyle: Diet and Bevicizumab+CM | Lifestyle: Diet+Exericise and Bevicizumab+CM
Number analyzed (Participants) | 11 | 13
cases | 10 | 5

5. Secondary Outcome: Number of Serious Adverse Event (AE) of Lifestyle
Description: Exercise and/or dietary lifestyle interventions defined per protocol. The lifestyle intervention will be administered by telephone, supplemented with a participant workbook (Appendix 9 in protocol). Only Grade 3/4 AE (CTCAE v4) was reported.
Time Frame: Followed every 6 months for 7.5 years after study entry, or completion of final analysis, whichever comes first.
Measure: Number; unit: cases
Arm/Group | Lifestyle: Diet | Lifestyle: Diet+Exericise | Lifestyle: Diet and Bevicizumab+CM | Lifestyle: Diet+Exericise and Bevicizumab+CM
Number analyzed (Participants) | 13 | 13 | 11 | 13
cases | 2 | 4 | 14 | 8

6. Secondary Outcome: Change in Level of Fasting Insulin
Description: Change in level of fasting insulin from baseline at study entry to 6 months.
Time Frame: Baseline and 6 months
Population: data not collected due to early termination of the study.
Arm/Group | Lifestyle: Diet | Lifestyle: Diet+Exericise | Lifestyle: Diet and Bevicizumab+CM | Lifestyle: Diet+Exericise and Bevicizumab+CM
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Change in Body Weight
Description: data not collected due to early termination of the study.
Time Frame: Baseline and 6 months
Population: This outcome will not be analyzed because there is not enough power to draw a meaningful conclusion on estimates due to early termination of the study.
Arm/Group | Lifestyle: Diet | Lifestyle: Diet+Exericise | Lifestyle: Diet and Bevicizumab+CM | Lifestyle: Diet+Exericise and Bevicizumab+CM
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: Change in IGF-1
Description: Change in level of insulin-like growth factor -1 (IGF-1) from baseline at study entry to 6 months.
Time Frame: Baseline and 6 months
Population: Results are not provided because the small sample size potentially identifies participants.
Arm/Group | Lifestyle: Diet | Lifestyle: Diet+Exericise | Lifestyle: Diet and Bevicizumab+CM | Lifestyle: Diet+Exericise and Bevicizumab+CM
Number analyzed (Participants) | 0 | 0 | 0 | 0

9. Secondary Outcome: Changes in Diet and Physical Activity Upon Biomarkers
Description: To evaluate the impact of changes in diet and physical activity upon biomarkers associated with breast cancer risk and prognosis, including leptin, adiponectin, testosterone, estradiol and inflammatory mediators (including: TNF alpha, IL-1 beta, IL-2, IL-5, IL-6, IL-8, IL-10, and IL-12)
Time Frame: Participants will undergo a series of measures at baseline and 6- and 12-months after study enrollment to assess the impact of the telephone-based lifestyle interventions upon biomarkers
Population: data not collected due to early termination of the study.
Arm/Group | Lifestyle: Diet | Lifestyle: Diet+Exericise | Lifestyle: Diet and Bevicizumab+CM | Lifestyle: Diet+Exericise and Bevicizumab+CM
Number analyzed (Participants) | 0 | 0 | 0 | 0

10. Secondary Outcome: Changes in Physical Activity and Dietary Behaviors
Time Frame: Participants will undergo a series of measures at baseline and 6- and 12-months after study enrollment to assess the impact of the telephone-based lifestyle interventions upon physical activity
Population: data not collected due to early termination of the study.
Groups:
- Observation + Diet/Diet and Exercise: Patients in observation group will receive following diet or diet + exercise intervention.
  The dietary intervention focuses on the Food Pyramid, emphasizing diet that is low in fat and high in fruits, vegetables and fiber. The exercise intervention is comprised of a target physical activity goal of 180 minutes of moderate-intensity activity each week. Patients receive a series of 13 telephone calls over the course of one-year with a dedicated and trained counselor.
- Bevicizumab+CM: Bevicizumab: 15 mg/kg administered intravenously day 1 of a 3-week cycle for 6 months and day 1 of a 6 week cycle up to 2 years Cyclophosphamide: 50 mg orally each day of a 3-week cycle for 6 months Methotrexate: 2.5 mg orally twice daily of a 3-week cycle for 6 months Patients will receive diet or diet + exercise intervention.
Arm/Group | Observation + Diet/Diet and Exercise | Bevicizumab+CM
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Impact Upon Anthropometric Measures, Quality of Life and Fatigue
Time Frame: as for outcome 10
Population: data not collected due to early termination of the study.
Arm/Group | Observation + Diet/Diet and Exercise | Bevicizumab+CM
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Disease assessments occurred every 12 weeks on treatment and every 6 months in long-term follow-up up to 7.5 years.
Arm/Group | Lifestyle: Diet | Lifestyle: Diet+Exericise | Lifestyle: Diet and Bevicizumab+CM | Lifestyle: Diet+Exericise and Bevicizumab+CM
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13 | 0/11 | 3/13
Serious Adverse Events (participants affected / at risk) | 2/13 | 3/13 | 11/11 | 8/13
Other Adverse Events (participants affected / at risk) | 13/13 | 13/13 | 11/11 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lifestyle: Diet (N=13) | Lifestyle: Diet+Exericise (N=13) | Lifestyle: Diet and Bevicizumab+CM (N=11) | Lifestyle: Diet+Exericise and Bevicizumab+CM (N=13)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Wound infection (Infections and infestations) | 0 | 0 | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 2 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lifestyle: Diet (N=13) | Lifestyle: Diet+Exericise (N=13) | Lifestyle: Diet and Bevicizumab+CM (N=11) | Lifestyle: Diet+Exericise and Bevicizumab+CM (N=13)
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 3 | 2
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Cardiac disorders - Other, specify (Cardiac disorders) | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 1
Edema limbs (General disorders) | 1 | 1 | 2 | 2
Edema trunk (General disorders) | 1 | 0 | 0 | 0
Facial pain (General disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 4 | 5 | 7 | 7
Fever (General disorders) | 0 | 0 | 1 | 0
Localized edema (General disorders) | 0 | 1 | 0 | 0
Pain (General disorders) | 5 | 0 | 4 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Nail loss (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 4 | 1 | 2 | 5
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 2 | 2
Nausea (Gastrointestinal disorders) | 1 | 0 | 5 | 5
Stomach pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gallbladder pain (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Allergic reaction (Immune system disorders) | 0 | 0 | 1 | 1
Lung infection (Infections and infestations) | 1 | 0 | 0 | 0
Mucosal infection (Infections and infestations) | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 2
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 2
Wound infection (Infections and infestations) | 0 | 0 | 0 | 1
Infections and infestations - Other, specify (Infections and infestations) | 1 | 0 | 1 | 2
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Venous injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 3 | 3
Alkaline phosphatase increased (Investigations) | 1 | 1 | 2 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 4 | 3
Blood bilirubin increased (Investigations) | 1 | 1 | 1 | 0
INR increased (Investigations) | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 1 | 1
Weight gain (Investigations) | 1 | 0 | 0 | 0
Weight loss (Investigations) | 1 | 0 | 0 | 0
White blood cell decreased (Investigations) | 1 | 2 | 2 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0 | 4 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 0 | 4 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 3
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 2 | 2 | 5
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 2
Headache (Nervous system disorders) | 2 | 2 | 4 | 3
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 1
Neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 0 | 5 | 4
Nervous system disorders - Other, specify (Nervous system disorders) | 0 | 1 | 0 | 0
Eye disorders - Other, specify (Eye disorders) | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 1 | 3 | 1
Confusion (Psychiatric disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 4 | 2
Insomnia (Psychiatric disorders) | 1 | 1 | 5 | 2
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 6 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hematuria (Renal and urinary disorders) | 1 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1 | 1
Urinary frequency (Renal and urinary disorders) | 2 | 0 | 0 | 2
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 | 0 | 0 | 1
Breast pain (Reproductive system and breast disorders) | 0 | 2 | 0 | 0
Irregular menstruation (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 2 | 0
Vaginal dryness (Reproductive system and breast disorders) | 4 | 0 | 1 | 1
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 1 | 0 | 0 | 0
Hematoma (Vascular disorders) | 0 | 0 | 0 | 1
Hot flashes (Vascular disorders) | 7 | 4 | 5 | 2
Hypertension (Vascular disorders) | 1 | 1 | 3 | 6
Lymphedema (Vascular disorders) | 2 | 0 | 0 | 2
Thromboembolic event (Vascular disorders) | 0 | 0 | 1 | 0
Vascular disorders - Other, specify (Vascular disorders) | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
The study was terminated early due to slow accrual and therefore interpretation of results is limited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No